CLINICAL TRIAL: NCT05543421
Title: Transcranial Magnetic Stimulation in Patients With a Depressive Episode
Brief Title: Transcranial Magnetic Stimulation in Patients With a Depressive Episode - RCT Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SUBZ.C230.22.062.TMS.MDD
Record Dates: First submitted 2022-06-06; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-06

CONDITIONS: Major Depressive Disorder
Keywords: TMS; iTBS; MDD; RCT
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- rTMS active (Active Comparator)
  Interventions: Device: TMS
- rTMS sham (Sham Comparator)
  Interventions: Device: TMS
- iTBS active (Experimental)
  Interventions: Device: TMS
- iTBS sham (Sham Comparator)
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — rTMS (30sessions) or iTBS (40sessions)

SUMMARY:
The study is planned as a randomized, double-blind, active comparator-controlled and sham-controlled parallel trial, in which raters and participants will be blinded to the group selection. A total of 60 participants, meeting the eligibility criteria, will be enrolled in the study and divided randomly into 4 groups (2 experimental ones with active rTMS or iTBS and 2 controls with sham-placebo rTMS or iTBS stimaltions).

DETAILED DESCRIPTION:
The study is planned as a randomized, double-blind, active comparator-controlled and sham-controlled parallel trial, in which raters and participants will be blinded to the group selection. A total of 60 participants, meeting the eligibility criteria, will be enrolled in the study and divided randomly into 4 groups (2 experimental ones and 2 controls):

1. EG1 (N=20) rTMS stimulation (1 session daily per 30 days, 3000 pulses per session, session time = 37,5 minutes, 10Hz),
2. EG2 (N=20) iTBS stimulation (4 short sessions daily per 14 days, 600 pulses per session, session time=3 minutes, 50Hz),
3. CG1 (N=10) placebo (sham-coil) stimulation based on rTMS protocol,
4. CG2 (N=10) placebo (sham-coil) stimulation based on iTBS protocol. Efficacy will be analyzed on the intention-to-treat population, defined as participants who completed the baseline and at least one evaluation after rTMS intervention.

The following are the inclusion and exclusion criteria for the recruitment process:

The following stimulation protocols will be used to conduct research into the treatment of depressive disorders:

1. Stimulation with rTMS within the left hemisphere, in the dorsolateral prefrontal cortex, DLPFC (Dorsolateral prefrontal cortex). In the field of stimulation, a protocol based on FDA recommendations, so- called train stimulation (stimulation of a given frequency for a short period of time with longer breaks without stimulation) assuming the following stimulation parameters:

   * Magnetic field intensity: 120% of the initial excitability threshold for the motor cortex,
   * Frequency: 10 Hz for 4 seconds of stimulation,
   * Breaks in stimulation: 26 seconds,
   * Total number of stimulation pulses: 3000,
   * Duration of one session: 37.5 minutes,
   * Duration of therapy: from 4 to 6 weeks (sessions on days 1-5, break on days 6 and 7).
2. iTBS protocol in the left cerebral hemisphere, in the dorsolateral prefrontal cortex, DLPFC (Dorsolateral prefrontal cortex). Expected range of parameters:

   * Frequency: up to 50 Hz, Intensity: 80% excitability threshold for the motor cortex,
   * Breaks between pulse series: up to 10 seconds
   * Duration of a single session: from 20 to 190 seconds,
   * Duration of treatment: 40 sessions,
   * Total number of pulses in a session: 600, sessions a day: 4.
   * Duration of one session: 3 minutes,
   * Duration of therapy: 2 weeks (sessions on days 1-5, break on days 6 and 7).

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric diagnosis (F3X);
* Symptom severity - total score of the Hamilton Depression Scale a least 17
* Granting informed consent
* The possibility for the patient to ensure constant participation in individual sessions and clinical evaluations, in particular in terms of place of residence and travel options
* 18-70 years of age.

Exclusion Criteria:

* Contraindications to treatments using TMS
* Lack of informed consent from the patient
* Documented persistent lack of cooperation in treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of efficiency of rTMS and iTBS active stimulation Change from Baseline to END of stimulation regarded as reduction of symptoms measured in MADRS scale | END of stimulation
  Comparison of efficiency of rTMS and iTBS active stimulation from baseline to end of stimualion measured with MADRS. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
Comparison of efficiency of rTMS and iTBS active stimulation Change from Baseline to 3 months of follow up after end of stimulation regarded as reduction of symptoms measured in MADRS scale | 3 months after end of stimulation
  Comparison of efficiency of rTMS and iTBS active stimulation from baseline to 3 months follow up after end of stimualion measured with MADRS. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
Comparison of efficiency of rTMS and iTBS active stimulation Change from Baseline to END of stimulation regarded as reduction of symptoms measured in HAMD scale | END of stimulation
  Comparison of efficiency of rTMS and iTBS active stimulation from baseline to end of stimualion measured with HAMD. The HAMD is a 17-items scale, measuring depression severity, the overall score ranges from 0 to 60, higher score means more severe depression.
Comparison of efficiency of rTMS and iTBS active stimulation Change from Baseline to 3 months of follow up after end of stimulation regarded as reduction of symptoms measured in HAMD scale | 3 months after end of stimulation
  Comparison of efficiency of rTMS and iTBS active stimulation from baseline to 3 months follow up after end of stimualion measured with HAMD. The HAMD is a 17-items scale, measuring depression severity, the overall score ranges from 0 to 60, higher score means more severe depression.
Comparison of efficiency of rTMS active and rTMS sham-placebo stimulation Change from Baseline to END of stimulation regarded as reduction of symptoms measured in MADRS scale | END of stimulation
  Comparison of efficiency of rTMS active and rTMS sham placebo stimulation from baseline to end of stimulation measured with MADRS. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
Comparison of efficiency of rTMS active and rTMS sham placebo stimulation from baseline to end of stimulation measured with MADRS | 3 months after end of stimulation
  Comparison of efficiency of iTBS active and iTBS sham-placebo stimulation Change from Baseline to END of stimulation regarded as reduction of symptoms measured in MADRS scale. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.

CONTACTS AND LOCATIONS:
Locations (1):
- Wroclaw Medical Univeristy, Department of Psychiatry, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided